CLINICAL TRIAL: NCT06445972
Title: A Phase 1/2 Open-Label, Umbrella Platform Design Study to Evaluate the Safety and Efficacy of Investigational Agents in Combination With Standard of Care Treatments as the Second-Line Treatment of Participants With Advanced/Metastatic Gastroesophageal Adenocarcinoma: Substudy 06D
Brief Title: Substudy 06D: Combination Therapies in Second Line (2L) Gastroesophageal Adenocarcinoma (MK-3475-06D/Keymaker-U06)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3475-06D; 2023-509306-29-00 (Registry Identifier: EU CT); U1111-1299-8160 (Registry Identifier: UTN); MK-3475-06D (Other: MSD)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Gastroesophageal Junction; Gastroesophageal Adenocarcinoma; Esophageal Neoplasms; Esophageal Cancer
Keywords: Programmed Cell Death 1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Ramucirumab; Paclitaxel; patritumab deruxtecan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ramucirumab + Paclitaxel (Active Comparator): Participants receive ramucirumab at 8mg/kg via intravenous (IV) infusion on days 1 and 15 of each 4-week cycle for up to ~60 weeks plus paclitaxel at 80 mg/M^2 via IV infusion on Days 1, 8, and 15 of each 4-week cycle (3 weeks on and 1 week off) until discontinuation.
  Interventions: Biological: Ramucirumab; Drug: Paclitaxel
- Sacituzumab Tirumotecan + Paclitaxel (Experimental): Following a 28-day run-in with sacituzumab tirumotecan at 3 mg/kg and 4 mg/kg IV infusion on Days 1 and 15 of a 6-week cycle plus paclitaxel at 80 mg/M^2 IV infusion on days 1, 8 and 15 of a 4-week cycle, participants receive paclitaxel at 80 mg/M^2 IV infusion on days 1, 8, 15 of each 4-week cycle (3 weeks on and 1 week off) plus sacituzumab tirumotecan at selected dose IV infusion on days 1, 15, 29 of every 6-week cycle until discontinuation.
  Interventions: Drug: Paclitaxel; Biological: Sacituzumab Tirumotecan; Drug: Rescue Medications
- HER3-DXd + Ramucirumab (Experimental): Participants receive HER3-DXd via IV infusion on days 1 and 22 of each 6-week cycle plus ramucirumab at 8mg/kg via IV infusion on days 1 and 15 and 29 of each 6-week cycle until discontinuation.
  Interventions: Biological: Ramucirumab; Drug: Rescue Medications; Biological: HER3-DXd

INTERVENTIONS:
Biological: Ramucirumab — 8 mg/kg IV Infusion
  Arms: HER3-DXd + Ramucirumab; Ramucirumab + Paclitaxel
Drug: Paclitaxel — 80 mg/M^2 IV infusion
  Arms: Ramucirumab + Paclitaxel; Sacituzumab Tirumotecan + Paclitaxel
Biological: Sacituzumab Tirumotecan — 3 mg/kg or 4 mg/kg IV Infusion
  Other Names: MK-2870; SKB264; sac-TMT
  Arms: Sacituzumab Tirumotecan + Paclitaxel
Drug: Rescue Medications — Participants receive rescue medications according to each approved drug's product label. Recommended rescue medications for the Sacituzumab Tirumotecan + Paclitaxel arm include antihistamines (histamine-1 and histamine-2 receptor antagonists), acetaminophen or equivalent, dexamethasone or equivalent infusion, and steroid mouth wash (dexamethasone or equivalent) and rescue medications for the HER3-DXd + ramucirumab arm include 5-HT3-receptor antagonist, NK-1 receptor antagonist, and corticosteroids.
  Arms: HER3-DXd + Ramucirumab; Sacituzumab Tirumotecan + Paclitaxel
Biological: HER3-DXd — IV Infusion
  Other Names: patritumab deruxtecan; MK-1022; U3-1402
  Arms: HER3-DXd + Ramucirumab

SUMMARY:
This is a phase 1/2 multicenter, open-label umbrella platform study that will evaluate the safety and efficacy of sacituzumab tirumotecan (MK-2870) plus paclitaxel versus ramucirumab plus paclitaxel, and HER3-DXD plus ramucirumab versus ramucirumab plus paclitaxel for the treatment of participants with advanced or metastatic gastric adenocarcinoma, gastroesophageal junction (GEJ) adenocarcinoma, or esophageal adenocarcinoma who have failed 1 prior line of therapy. This is an estimation study, and no formal hypothesis testing will be performed.

DETAILED DESCRIPTION:
This is a substudy of the master protocol MK-3475-U06 (KEYMAKER-U06).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically and/or cytologically confirmed diagnosis of previously treated, second line (2L) (received first line (1L) treatment) gastric adenocarcinoma, gastroesophageal junction adenocarcinoma, or esophageal adenocarcinoma
* Has metastatic disease or locally advanced, unresectable disease
* Has experienced documented objective radiographic or clinical disease progression during or after 1L therapy containing any platinum/fluoropyrimidine doublet with or without immunotherapy
* Tumor tissue must be confirmed as negative for HER2 expression (IHC 0/1+ or IHC2+/in situ hybridization negative) as classified by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines
* Can provide a core/excisional biopsy of a tumor lesion not previously irradiated (collected from a biopsy performed after the most recent systemic anticancer therapy regimen)
* AEs due to previous anticancer therapies must be ≤Grade 1 or baseline (except alopecia and vitiligo). Endocrine-related AEs adequately treated with hormone replacement are acceptable
* Has Eastern Cooperative Oncology Group performance status of 0 or 1
* Has a life expectancy of at least 3 months
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to allocation/randomization
* Participants with history of Hepatitis C Virus (HCV) infection are eligible if HCV viral load is undetectable at screening
* Human Immunodeficiency Virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has squamous cell or undifferentiated gastroesophageal cancer
* Has experienced weight loss >20% over 3 months before the first dose of study intervention
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has Grade ≥2 peripheral neuropathy
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has a serious or nonhealing wound or peptic ulcer or bone fracture within 28 days prior to allocation/randomization
* Has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (hemicolectomy or extensive small intestine resection with chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Has experienced any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to allocation/randomization
* Has uncontrolled arterial hypertension ≥150/≥90 mm mercury (Hg)
* Has accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks prior to enrollment
* Has undergone major surgery within 28 days prior to allocation/randomization, or central venous access device placement within 7 days prior to allocation/randomization or planned major surgery following initiation of study treatment
* Is receiving therapeutic anticoagulation with warfarin, low-molecular weight heparin or similar agents
* Is receiving chronic therapy with nonsteroidal anti-inflammatory agents or other antiplatelet agents
* Has a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism during the 3 months prior to allocation/randomization
* Has significant bleeding disorders, vasculitis, or had a significant bleeding episode from the gastrointestinal (GI) tract within 3 months prior to study entry
* Has history of GI perforation and/or fistulae within 6 months prior to allocation/randomization
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has received prior treatment with a trophoblast cell-surface antigen 2 (TROP2)- or HER3-targeted agent, topoisomerase 1 inhibitor-based ADC and/or a topoisomerase 1 inhibitor-based chemotherapy, or any previous systemic therapy targeting vascular endothelial growth factor (VEGF) or the vascular endothelial growth factor receptor (VEGFR) signaling pathways
* Has received prior systemic anticancer therapy within 4 weeks before the first dose of study intervention
* Has received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years. Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded
* Has known active central nervous system metastases and/or carcinomatous meningitis
* Has an active infection requiring systemic therapy
* Has concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV deoxyribonucleic acid) and Hepatitis C virus (defined as anti-HCV antibody positive and detectable HCV ribonucleic acid) infection
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease, or where suspected ILD or pneumonitis cannot be ruled out by imaging at screening
* Has severe hypersensitivity (Grade ≥3) to MK-2870, or HER3-DXd, any of their excipients, and/or to another biologic therapy
* Has not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2030-10-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Experience Dose Limiting Toxicities (DLTs) During the Safety Lead-In Phase | Up to ~28 days
  DLTs are defined as any drug-related adverse event (AE) according to the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) Version 5.0, observed during the DLT evaluation period that results in a change to a given dose or a delay in initiating the next cycle. The percentage of participants who experience at least one DLT will be presented.
Percentage of Particiapants who Experience an Adverse Event (AE) During the Safety Lead-In Phase | Up to ~60 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued study intervention due to an AE will be presented.
Percentage of Participants who Discontinue Study Intervention Due to an AE During the Safety Lead-In Phase | Up to ~28 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued study intervention due to an AE will be presented.
Objective Response Rate (ORR) | Up to ~28 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to ~50 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Duration of Response (DOR) | Up to ~50 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Overall Survival (OS) | Up to ~50 months
  OS is defined as the time from the date of randomization to the date of death from any cause. OS will be presented.
Percentage of Particiapants who Experience an AE During the Efficacy Phase | Up to ~50 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued study intervention due to an AE will be presented.
Percentage of Participants who Discontinue Study Intervention Due to an AE During the Efficacy Phase | Up to ~50 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued study intervention due to an AE will be presented.
Incidence of sacituzumab tirumotecan anti-drug antibody (ADA) | Up to ~50 months
  In participants treated with sacituzumab tirumotecan the immunogenicity of sacituzumab tirumotecan ADA response will be evaluated with validated immunogenicity assays.
Incidence of HER3-DXd ADA | Up to ~50 months
  In participants treated with HER3-DXd, the immunogenicity of HER3-DXd ADA response will be evaluated with validated immunogenicity assays.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (42):
- United States (8):
  - University of Arizona Cancer Center-University of Arizona Cancer Center ( Site 8927), Tucson, Arizona
  - UCLA Hematology/Oncology - Santa Monica ( Site 8905), Los Angeles, California
  - Norton Cancer Institute - Downtown ( Site 8900), Louisville, Kentucky
  - The Cancer and Hematology Centers ( Site 8912), Grand Rapids, Michigan
  - Hematology-Oncology Associates of Central NY, P.C. ( Site 8925), East Syracuse, New York
  - Columbia University Irving Medical Center-CUIMC Herbert Irving Comprehensive Cancer Center Clinical ( Site 8907), New York, New York
  - UPMC Hillman Cancer Center-UPMC ( Site 8904), Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center ( Site 8920), Houston, Texas
- Brazil (3):
  - Liga Norte Riograndense Contra o Câncer ( Site 8303), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceição ( Site 8301), Porto Alegre, Rio Grande do Sul
  - IBCC - Instituto Brasileiro de Controle do Câncer ( Site 8304), São Paulo, São Paulo
- Chile (7):
  - Clínica Puerto Montt ( Site 8409), Port Montt, Los Lagos Region
  - Centro de Investigación del Maule ( Site 8408), Talca, Maule Region
  - FALP-UIDO ( Site 8400), Santiago, Region M. de Santiago
  - Centro de Oncología de Precisión-Oncology ( Site 8404), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo ( Site 8405), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 8401), Santiago, Region M. de Santiago
  - Bradford Hill Norte ( Site 8407), Antofagasta
- China (8):
  - Beijing Cancer hospital-Digestive Oncology ( Site 7500), Beijing, Beijing Municipality
  - The 900th Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army ( Site 7501), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 7503), Xiamen, Fujian
  - Henan Cancer Hospital ( Site 7504), Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University ( Site 7514), Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center ( Site 7513), Shanghai, Shanghai Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi ( Site 7506), Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine ( Site 7510), Hangzhou, Zhejiang
- France (3):
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital-Institut de cancérologie et hématologi ( Site 7104), Brest, Finistere
  - CIC. ( Site 7100), Lille, Nord
  - Pitie Salpetriere University Hospital-Hepato-Gastro-Enterology ( Site 7102), Paris, Île-de-France Region
- Germany (2):
  - Universitaetsklinikum Duesseldorf-Gastroenterology, Hepatology and Infectiology ( Site 8802), Düsseldorf, North Rhine-Westphalia
  - Facharztzentrum Eppendorf-Facharztzentrum Eppendorf ( Site 8807), Hamburg
- Italy (2):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori"-Oncologia Medica ( Site 7207), Meldola, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 7200), Milan, Lombardy
- Oslo universitetssykehus, Radiumhospitalet ( Site 8501), Oslo, Norway
- South Korea (2):
  - Asan Medical Center-Department of Oncology ( Site 7901), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 7900), Seoul
- Switzerland (2):
  - Hôpitaux Universitaires de Genève (HUG) ( Site 8701), Geneva, Canton of Geneva
  - Kantonsspital Graubünden-Medizin ( Site 8700), Chur, Kanton Graubünden
- Taiwan (4):
  - China Medical University Hospital ( Site 8007), Taichung
  - National Cheng Kung University Hospital ( Site 8001), Tainan
  - National Taiwan University Hospital-Oncology ( Site 8000), Taipei
  - Taipei Veterans General Hospital ( Site 8005), Taipei

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26286&tenant=MT_MSD_9011